CLINICAL TRIAL: NCT04993170
Title: Systematic Analysis of a Standardized Questionnaire to Detect Possible Bleeding Disorders Used in Clinical Routine During Anaesthesiological Preoperative Assessment and Its Impact on Perioperative Hemostasis Management
Brief Title: Systematic Analysis of a Standardized Questionnaire to Detect Possible Bleeding Disorders and Its Impact on Perioperative Hemostasis Management
Acronym: PrEdict
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Institute for biometry and clinical epidemiology, Charité University Berlin, Germany (Unknown); Institute for transfusion medicine, Charité University Berlin, Germany (Unknown); Einstein center digital future (Unknown)
Responsible Party: Principal Investigator, Sascha Treskatsch, Univ.-Prof. Dr. med., Head of Department, Charite University, Berlin, Germany
Other Study IDs: EA4/181/20
Record Dates: First submitted 2021-07-05; First posted 2021-08-06 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Perioperative Hemorrhage; Hemostasis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Bleeding assessment tool — The standardized application of the questionnaire serves to identify patients at risk of bleeding at an early stage and to adapt and optimize perioperative coagulation management accordingly by initiating targeted diagnostics and therapy

SUMMARY:
With the help of a standardized questionnaire, an increased risk of bleeding due to pre-existing hemostasis disorders in the site-specific patient population will be detected and the corresponding enhanced diagnostic measures will be initiated. The planned prospective observational study should i.) systematically investigate the results of this procedure and ii.) allow a comparison with a retrospective perioperative cohort that was cared for at the Benjamin Franklin Campus before the introduction of the questionnaire. Due to the campus structure with a large vascular surgery center as well as a large urological, general and trauma surgery department, a high number of multimorbid patients with pre-existing disorders of primary hemostasis, mainly caused by medication or secondary diseases, is to be expected.

In the following, the feasibility of the required measures in clinical routine (measured by the frequency of actual changes or modifications of the initially planned perioperative procedure, the adequate implementation of indicated diagnostic measures, etc.) will be examined.

DETAILED DESCRIPTION:
The aim of the study is the systematic scientific evaluation of a standardized questionnaire for bleeding history already used in clinical routine during the preoperative anesthesiological visit and its impact on perioperative coagulation management.

The routine use of a standardized questionnaire to assess bleeding risk is based on a study on the preoperative identification of patients with (primary) hemostasis disorders from 2007: in a patient collective of 5649 patients from different disciplines at the Charité - Universitätsmedizin Berlin, a positive predictive value of 99% for the presence of a hemostasis disorder could be established if at least four questions of a standardized bleeding history questionnaire were answered positively. This is not possible in the same way with the plasmatic coagulation-global tests established in clinical routine.

The standardized application of the questionnaire serves to identify patients at risk of bleeding at an early stage and to adapt and optimize perioperative coagulation management accordingly by initiating targeted diagnostics and therapy. However, a systematic scientific evaluation of this questionnaire with regard to the conditions at the Benjamin Franklin Campus with a large vascular surgery center as well as a large urological, general and trauma surgery department and a high number of multimorbid patients with pre-existing disorders of primary hemostasis, mainly caused by medication or secondary diseases, is still pending.

ELIGIBILITY:
Inclusion Criteria:

All adult (age ≥ 18 years) patients of both genders undergoing elective surgery at the Benjamin Franklin campus in the 12-month period

Exclusion Criteria:

* Pregnancy, lactation
* Patients not capable of giving consent
* Already diagnosed hemostasis disorder
* Patients under (plasmatic) anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult (age ≥ 18 years) patients of both sexes undergoing elective surgery at the Benjamin Franklin Campus in the period of 12 months and presenting at the anesthesiological preoperative assessment will be recorded.
  A historical cohort that received surgical care at the Benjamin Franklin campus prior to the introduction of the questionnaire (07/01/2018 - 06/30/2019) will serve as the comparison group.
Sampling Method: Non-Probability Sample
Enrollment: 5004 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Relative frequency of changes in the initially planned perioperative procedure | Perioperative period
  The relative frequency of changes in the initially planned perioperative procedure in patients with abnormalities in the preoperative questionnaire and target-oriented laboratory diagnostics will be measured.
  Changes can be:
  * need for extended coagulation diagnostics
  * hemostaseological consultation preoperatively
  * administration of coagulation-active substances

SECONDARY OUTCOMES:
Perioperative complications | Perioperative period
  Compared to a retrospective control group in which no standardized questionnaire was used, the use of a standardized questionnaire and the targeted diagnostics initiated in case of abnormalities lead to
  * lower blood loss (estimated in ml, qualitatively)
  * a lower transfusion rate during surgery (number of red cell concentrates)
  * less time spent in the recovery room (hours:minutes)
  * a lower rate of revision surgery due to postoperative bleeding (number of patients)
  * fewer organ complications (number of patients, organ failure defined and diagnosed by attending physician)
Diagnostic discrepancy | Perioperative period
  There is a discrepancy between the number of patients, for whom additional diagnostics and measures ,based on the evaluation of the questionnaire,are required on the one hand, and the number ob patients, fo whom these additional diagnostics and measures are actually performed at the time of surgery on the other hand. The relative frequency of these discrepancies should be determined.
  Additional diagnostics and measures are:
  * extended coagulation diagnostics
  * hemostaseological consultation preoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Campus Benjamin Franklin, Charité - Universitätsmedizin Berlin, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: No